CLINICAL TRIAL: NCT01064947
Title: Use of Altabax Ointment (Retapamulin 1%) BID for 7 Days in Treatment of Secondary Infection With Staphylococcus Aureus (MRSA and MSSA) and Streptococcus Pyogenes in Atopic Dermatitis Patients - Open Label Pilot Study
Brief Title: Safety and Efficacy Study of Altabax Ointment in the Treatment of Secondarily Infected Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Leon Kircik, M.D., Principal Investigator, Derm Research, PLLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALT113706
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2013-04

CONDITIONS: Atopic Dermatitis; Secondary Infection
MeSH Terms: conditions — Dermatitis, Atopic; Coinfection | interventions — retapamulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Retapamulin 1% — Apply a thin layer of Retapamulin 1% to the affected area twice daily. The treated area may be covered with a sterile bandage or gauze dressing if desired.
  Other Names: Altabax

SUMMARY:
Skin infections may complicate the treatment of atopic dermatitis.The use of topical ointments has become very important to avoid the use of oral antibiotics. There is little supporting literature regarding the use of topical antibiotics in secondarily infected atopic dermatitis.

This study will investigate the safety and effectiveness of Altabax ointment use in treating secondarily infected atopic dermatitis caused by Staphylococcus aureus and Streptococcus pyogenes.

DETAILED DESCRIPTION:
Atopic dermatitis patients are commonly secondarily infected with Staphylococcus aureus and/or Streptococcus pyogenes, more recently with Methicillin-resistant Staphylococcus aureus (MRSA), due to impaired barrier function. As cutaneous infections such as MRSA and others may complicate the treatment of atopic dermatitis, the use of topical antibiotics have become very important to avoid oral antibiotics and their side effects, especially in the pediatric population.

The current study will investigate the safety and efficacy of Altabax ointment use for treatment of secondarily infected lesions caused by Staphylococcus aureus and Streptococcus pyogenes in both the pediatric and adult populations.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of childbearing potential must have a negative urine pregnancy test at Baseline and practice a reliable method of contraception.
* Secondary infection of atopic dermatitis with S.aureus or S.pyogenes as the probable causative agent.
* An infected area less than or equal to 100 centimeters squared for subjects 18 years of age or older, or, 2% body surface area for subjects under 18 years of age.
* Skin Infection Rating Scale score greater than or equal to 8.
* Able to understand and comply with the requirements of the study and sign Informed Consent/Health Insurance Portability and Accountability Authorization Forms. Subjects under the legal age of consent must also have the written informed consent of parent or legal guardian.

Exclusion Criteria:

* Female subjects who are pregnant, trying to get pregnant, breast feeding or who are of childbearing potential and not practicing reliable birth control.
* Allergic to any component of the test medication.
* Clinical diagnosis of impetigo, folliculitis or minor soft tissue infection.
* Use of topical antibacterial medication to the study treatment area within 1 day of Visit 1.
* Signs of systemic infection or evidence of abcess or cellulitis at the site to be treated.
* Medical condition that,in the opinion of the investigator, contraindicates the subject's participation in the clinical study.
* Recent alcohol or drug abuse is evident.
* History of poor cooperation, non-compliance with medical treatment or unreliability.
* Participation in an investigational drug study within 30 days of Baseline Visit.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H. Kircik, M.D., Principal Investigator — DermResearch, PLLC
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with suspected secondarily infected atopic dermatitis were recruited from the investigator's medical practice. Recruitment occurred from July 2010 through November 2011
Pre-assignment Details: Seventy subjects were enrolled into the study. Of these 29 had a positive culture for s. aureus (MRSA and MSSA) or S. pyogenes
Groups:
- All Participants: All consented subjects with an apparent secondary infection were cultured.The treatment of Retapamulin 1% was started , with a thin layer applied twice daily and covered with gauze (if desired) for 7 days. The subject treatment site was cultured after 7 days of treatment.
Period: Overall Study
Arm/Group | All Participants
Started | 70
Completed | 29
Not Completed | 41
Not completed — negative culture | 41

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided only for those subjects with a positive culture
Groups:
- All Participants: All consented subjects with a suspected secondary infection of atopic dermatitis were cultured.The treatment of Retapamulin 1% was started , with a thin layer applied twice daily and covered with gauze (if desired) for 7 days. The subject treatment site was cultured after 7 days of treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 36.6 [2.1 to 76.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Bacteriological Culture
Description: All participants were cultured for S.aureus (MRSA), S.aureus (MSSA) and S. pyogenes at Baseline. If positive at Baseline then they were cultured again at Day 7.
Time Frame: Day 1 and Day 7
Measure: Number; unit: participants
Groups:
- All Participants at Day 1: All consented subjects with an apparent secondary infection were cultured.The treatment of Retapamulin 1% was started , with a thin layer applied twice daily and covered with gauze (if necessary) for 7 days. The subject treatment site was cultured after 7 days of treatment.
Arm/Group | All Participants at Day 1 | Participants With a Positive Culture at Day 1
Number analyzed (Participants) | 70 | 29
participants
  S. aureus (MRSA) | 13 | 3
  S. aureus (MSSA) | 16 | 5
  S. pyogenes | 0 | 0

2. Secondary Outcome: Skin Infection Rating Scale (SIRS)
Description: The Primary Investigator rated the each of the following characteristics: exudate/pus, crusting, erythema/inflammation, tissue warmth, tissue edema, itching and pain on a scale of 0-6 (absent-severe) to create an overall SIRS score ranging from 0-42.
Time Frame: Day 1 and Day 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Participants With Positive Culture at Day 1
Number analyzed (Participants) | 29
units on a scale
  SIRS at Day 1 | 10.0 [9.0 to 12.0]
  SIRS at Day 7 | 1.0 [1.0 to 3.0]

3. Secondary Outcome: Investigator Assessment of Clinical Cure
Description: The investigator assessed clinical cure at Day 7 as either total or improved cure, failure confirmed or failure by default
Time Frame: Day 7
Measure: Number; unit: participants
Arm/Group | Participants With a Positive Culture at Day 1
Number analyzed (Participants) | 29
participants
  clinical cure total | 12
  clinical cure improved | 15
  failure - confirmed and default | 2

4. Secondary Outcome: Local Tolerability
Description: The investigator assessed the following characteristics on a grading scale of 0-3 (none, mild moderate or severe): erythema, inflammation, infection, crusting, necrosis, peeling, swelling and contact dermatitis.
  The subject assessed the following characteristics on a scale of 0-3 (none, mild, moderate or severe): irritation, itchiness burning, tenderness and pain.
Time Frame: Day 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 29
units on a scale
  erythema | 1.00 [0.00 to 1.00]
  crusting | 0.00 [0.00 to 1.00]
  necrosis | 0.00 [0.00 to 0.00]
  inflammation | 0.00 [0.00 to 0.00]
  swelling | 0.00 [0.00 to 0.00]
  infection | 0.00 [0.00 to 0.00]
  peeling | 0.00 [0.00 to 0.00]
  contact dermatitis | 0.00 [0.00 to 0.00]
  iritation | 0.00 [0.00 to 0.00]
  itchiness | 0.00 [0.00 to 1.00]
  burning | 0.00 [0.00 to 0.00]
  tenderness | 0.00 [0.00 to 0.00]
  pain | 0.00 [0.00 to 0.00]

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

LIMITATIONS AND CAVEATS:
small number of subjects/short duration of study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No